CLINICAL TRIAL: NCT01770418
Title: A Phase I/II Study of Hypofractionated Proton Therapy for Stage II-III Non-Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Proton Collaborative Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUN005-12
Record Dates: First submitted 2013-01-11; First posted 2013-01-17 (Estimated); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Lung Neoplasms
Keywords: Non Small Cell Lung Cancer; Cancer; Lung; Proton; Radiation
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Proton Radiotherapy with Chemotherapy (Experimental)
  Interventions: Radiation: Radiation with Concurrent Chemotherapy

INTERVENTIONS:
Radiation: Radiation with Concurrent Chemotherapy — RADIATION: Proton Radiotherapy
  Dose Level 1: 60 Gy (RBE) at 2.5 Gy(RBE) per fraction x 24 fractions
  Dose Level 2: 60 Gy (RBE) at 3 Gy (RBE) per fraction x 20 fractions
  Dose Level 3: 60.01 Gy (RBE) at 3.53 Gy (RBE) per fraction x 17 fractions
  Dose Level 4: 60 Gy (RBE) at 4 Gy (RBE) per fraction x 15 fractions
  CONCURRENT CHEMOTHERAPY:
  Paclitaxel at a dose of 45 mg/m2 and Carboplatin at a dose of AUC 2 mg/min/ml (a total of 3-5 weekly doses) OR Cisplatin 50mg/m2 days 1, 8, 29, and 36 and Etoposide 50mg/m2 days 1-5, 29-33. For non squamous histology, Carboplatin AUC 5 on day 1 and Pemetrexed 500 mg/m2 on day 1 every 21 days OR Cisplatin 75 mg/m2 on day 1 and Pemetrexed 500 mg/m2 on day 1 every 21 days.
  Adjuvant chemotherapy is optional.

SUMMARY:
The purpose of this research study is to compare the effects (good and bad) on subjects and their cancer using standard chemotherapy in combination with hypofractionated proton radiation therapy. Hypofractionation is a technique that delivers higher daily doses of radiation over a shorter period of time.

DETAILED DESCRIPTION:
Conventional fractionated photon-based radiotherapy to 60-63 Gy at 1.8-2 Gy/fraction with concurrent chemotherapy remains the standard treatment practice in patients with stage III non-small cell lung carcinoma (NSCLC) with local control rates of approximately 50% and a median overall survival of just 18 months.Unfortunately, even the standard treatment has significant toxicity with approximately 40% of patients developing grade 3 or higher acute toxicities in the RTOG 9410 study.1 These outcomes are poor and more effective treatment regimens are needed.

Higher doses of radiation have been hypothesized to improve local control in patients with stage III NSCLC. This is expected to translate into better overall survival.Given the significant improvements in outcome in patients receiving hypofractionation for stage I NSCLC, perhaps similar gains could be achieved if hypofractionated radiotherapy could be safely delivered to stage II-III NSCLC with concurrent chemotherapy. Hypofractionated radiotherapy may offer improvement in local control compared with conventional fractionation that may translate into improved overall survival. Furthermore, hypofractionation will shorten the time interval during which patients are receiving less aggressive chemotherapy. Proton therapy is a highly conformal radiotherapy technique that takes advantage of the proton's characteristic Bragg Peak, resulting in significant reductions in the exit dose of the treatment beam. Thus, proton therapy can substantially reduce the dose to critical structures even compared with IMRT.

This study will investigate the safety and efficacy of delivering hypofractionated proton therapy with concurrent chemotherapy in patients with stage II-III NSCLC

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed invasive non-small cell lung cancer within 12 weeks prior to study registration. OR Pathologically confirmed invasive non-small cell lung cancer within 6 months prior to study registration if the patient received induction chemotherapy.
* AJCC (American Joint Committee on Cancer) 7th Ed. clinical stage II-III.
* ECOG Performance status 0-1 within 8 weeks prior to study registration.
* Patient must give study-specific informed consent on an IRB-approved consent prior to any research-related procedures or study treatment.
* Patient must be at least 18 years old at the time of consent.
* Patient must complete all required tests in section 4.
* Lab results per the following within 4 weeks prior to study registration:

  * Absolute neutrophil count (ANC) >1,800 cells/mm3.
  * Platelets > = 100,000 cells/mm3.
  * Hemoglobin > =10 g/dl. The use of transfusion or other intervention to achieve Hgb ≥10.0 g/dl is acceptable.
  * AST/SGOT and ALT/SGPT < 2.5 x the institutional upper limit of normal (IULN).
* Post exploratory thoracotomy must be done > 3 weeks prior to study registration or patient did not have post exploratory thoracotomy.
* PFT (pulmonary function test) with a FEV1 > 0.75 liters/second within 16 weeks prior to study registration.
* Patients must be evaluated by a thoracic surgeon, pulmonologist or medical oncologist and deemed medically or surgically unacceptable for resection.

Exclusion Criteria:

* Evidence of distant metastasis (M1) involvement.
* Prior radiotherapy to thoracic area.
* Unintentional weight loss >10% within 4 weeks prior to study registration.
* Pregnant and/or breast-feeding women, or patients (men and women) of child-producing potential not willing to use medically acceptable forms of contraception while on study treatment and for at least 12 months after study treatment. Pregnancy testing is not necessary for women who have had a hysterectomy or have not had a menstrual period for at least 24 consecutive months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-03; Primary Completion 2038-01 (Estimated)

PRIMARY OUTCOMES:
Phase I: Establish the maximum tolerated dose of radiotherapy in terms of Gy (RBE)/fraction using hypofractionated proton therapy concurrently with chemotherapy. | Weekly until completion of radiation treatment
  This phase will have a minimum of 2 treated patients and we anticipate that the MTD will be located before a maximum of 28 patients are treated. The trial begins by treating 5 patients at 2.5 Gy (RBE)/fraction to a dose of 60 Gy (RBE).
Phase II: Determine the percentage of patients that survive at least 12 months | At 12 months

SECONDARY OUTCOMES:
Assess acute and late adverse events of concurrent chemotherapy with hypofractionated proton therapy. | On average every 3 months for 5 years
Analyze for disease control and overall survival. | At 2 years and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Brad Hoppe, MD, Study Chair — Proton Collaborative Group
Locations (6):
- United States (6):
  - University of Florida Proton Therapy Institute, Jacksonville, Florida
  - Northwestern Medicine Chicago Proton Center, Warrenville, Illinois
  - Maryland Proton Treatment Center, Baltimore, Maryland
  - Princeton ProCure Management LLC, Somerset, New Jersey
  - Oklahoma Proton Center, Oklahoma City, Oklahoma
  - Hampton University Proton Therapy Institute, Hampton, Virginia